CLINICAL TRIAL: NCT03734055
Title: Peer Approaches to Lupus Self-management
Acronym: PALS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00080875; 1R01NR017892-01A1 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-11-07 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus; Quality of Life; Behavior, Health
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Health Behavior | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer Mentoring (Experimental): The program will consist of 12 sessions of peer mentoring that will include one standard educational session by telephone or video for approximately 60 minutes every 2 weeks. Additional interaction will be discouraged, but mentees and mentors will be asked to report any additional social interaction should it occur. The bi-weekly educational session will be generally structured in three parts: introduction, structured education, and problem solving. 60-minute calls are necessary for the delivery of educational content and mentors and mentees to be able to discuss their own experiences and potential solutions.
  Interventions: Behavioral: Peer Mentoring
- Social Support Group (Active Comparator): Mentees randomized to the social support control group will be enrolled in a lupus support group designed specifically for this project.
  Interventions: Behavioral: Social Support Group
- Peer Mentors (No Intervention): The principal roles of the peer mentors are to: 1) provide information about SLE, SLE-related behaviors, thoughts, and feelings, and the nature of recommended treatments; 2) provide social support to alleviate the mentee's sense of social isolation; 3) enhance and reinforce the mentee's sense of self-efficacy to manage their condition; and 4) encourage the mentee to participate actively in the recommended self-management skills building therapy.

INTERVENTIONS:
Behavioral: Peer Mentoring — Manualized peer mentorship program designed to provide modeling and reinforcement by peers (mentors) to other African American women with SLE (mentees) to encourage them to engage in activities that promote disease self-management.
  Arms: Peer Mentoring
Behavioral: Social Support Group — Social support controls will participate in a lupus support group created for this project, on the same schedule as peer mentoring sessions.
  Arms: Social Support Group

SUMMARY:
The Peer Approaches to Lupus Self-Management (PALS) study is a randomized, controlled in which 360 African American women with lupus will be recruited from the MUSC SLE database (60 mentors and 300 mentees). The peer mentoring intervention (patients will be matched with peer mentors who are considered competent in the management of their condition to provide modeling and reinforcement to participants) will occur by telephone for approximately 60 minutes every two weeks for 24 weeks. All participants will be assessed at baseline, mid-intervention (12 weeks post-enrollment), immediately following the intervention (24 weeks post-enrollment), and 12 months post-enrollment. The study will last 60 months with recruitment and enrollment over 48 months, 6 months for intervention delivery and 6 months for data analysis.

DETAILED DESCRIPTION:
The Peer Approaches to Lupus Self-Management (PALS) study is a randomized controlled trial designed to examine whether a new, culturally tailored peer mentoring intervention improves disease self-management, indicators of disease activity, and health related quality of life (HRQOL) in African American women with systemic lupus erythematosus (SLE). African American women with active SLE will be recruited as mentees and peer mentors. The investigators will recruit 300 mentees (150 mentored and 150 support group) and up to 60 mentors. As part of each wave, mentors (n=20) will be trained to deliver intervention content, prior to being paired with up to three mentees (n=50). The peer mentoring intervention will occur by twelve 60-minute telephone or video sessions carried out across the course of 24 weeks. In each wave, social support controls (n=50) will participate in a lupus support group created for this project, on the same schedule as peer mentoring sessions. Both conditions will be delivered via Webex, which has several advantages for this intervetion: 1) Sessions are easily accesible via phone or computer, allowing participants to choose their preferred interaction style; 2) A study coordinator can host the support groups and drop in/out for monitoring purposes; 3) There are video- or voice-call options for up to 25 paricipants at a time; and 4) This application ensures concordiant delivery methods across both arms of the study and the ability to document the frequency that voice and video options are used to adjust for participant choices in analyses. All participants (mentees, mentors, and social support controls) will be assessed using validated measures of patient reported outcomes and clinical indicators of disease activity at baseline, mid-intervention (3 months from baseline), immediately post-intervention (6 months from baseline), and 6 months post-intervention (12 months from baseline). For each wave, outcomes for mentees randomized to the mentored group will be compared with the outcomes of mentees randomized to the support group. A booster session will be incorporated for all participants (mentored and support group) at 3 months post-intervention to encourage retention.

ELIGIBILITY:
Inclusion Criteria:

* African American race/ethnicity
* Female sex
* Clinical diagnosis of SLE from a physician, according to ACR revised criteria for SLE
* 18 years of age or older

Additional inclusion criteria for mentors include:

* Disease duration > 2 years
* Able to attend scheduled training sessions
* Willing to provide one-on-one support to up to three African American women with SLE

Exclusion Criteria:

* Mentees who participated in the pilot will be ineligible to participate in this study as a mentee, but could participate as a mentor if they meet other eligibility criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Williams, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available. All findings will be reported in aggregate terms.

REFERENCES:
- [Derived] Leung J, Keller EP, Nietert P, Caldwell T, Dismuke-Greer CL, Johnson H, Williams E. Does social support reduce bodily pain among African American women with SLE? Findings from a randomised controlled trial. Lupus Sci Med. 2025 Oct 20;12(2):e001712. doi: 10.1136/lupus-2025-001712. PMID 41120192
- [Derived] Williams EM, Egede L, Oates JC, Dismuke CL, Ramakrishnan V, Faith TD, Johnson H, Rose J. Peer approaches to self-management (PALS): comparing a peer mentoring approach for disease self-management in African American women with lupus with a social support control: study protocol for a randomized controlled trial. Trials. 2019 Aug 23;20(1):529. doi: 10.1186/s13063-019-3580-4. PMID 31443732

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Mentoring | Social Support Group
Started | 182 | 132
Mentors | 44 | 0
Mentees | 138 | 132
Completed | 161 (Mentors Completed: 39 (5 Not Completed) Mentees Completed: 122 (16 Not Completed)) | 129
Not Completed | 21 | 3

BASELINE CHARACTERISTICS:
Population: Peer mentors administered the peer mentoring intervention and were not involved in social support groups.
Groups:
- Mentors: Peer mentors administered the peer mentoring intervention and were not involved in social support groups.
- Total: Total of all reporting groups
Arm/Group | Peer Mentoring | Social Support Group | Mentors | Total
Number analyzed (Participants) | 138 | 132 | 44 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (2.82) | 48 (2.82) | 49 (2.82) | 47 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 132 | 44 | 314
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 138 | 132 | 44 | 314
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 138 | 132 | 44 | 314
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 138 | 132 | 44 | 314

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction in Quality of Life as Assessed by the LUP-QOL (Lupus Quality of Life Questionnaire
Description: Quality of life will be assessed by using The LUP-QOL (Lupus Quality of Life Questionnaire), which assesses areas of the participant's life that may be affected by lupus. The score ranges from 0-100. A score of '0' indicates the lowest quality of life, and a score of 100 indicates the best quality of life. The 'Overall Impact' field reported has a scale of 0-700. Higher values represent a better outcome.
Time Frame: Baseline to 12 months post-intervention
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Mentoring | Social Support Group
Number analyzed (Participants) | 122 | 129
units on a scale | 330.50 (15.76) | 332.34 (15.75)

2. Primary Outcome: Change in Self-management
Description: The Patient Activation Measure (PAM) assesses an individual's knowledge, skill, and confidence for managing their health and healthcare. Individuals who measure high on this assessment typically understand the importance of taking a proactive role in managing their health and have the skills and confidence to do so. The PAM survey measures patients on a 0-100 scale and can segment patients into one of four activation levels along an empirically derived continuum, including "Believes Active Role Important", "Confidence and Knowledge to Take Action", "Taking Action", and "Staying Course Under Stress". Each activation level reveals insight into an array of health-related characteristics, including attitudes, motivators, behaviors, and outcomes. A high score represents a better outcome.
Time Frame: Baseline to 12 months post-intervention
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Mentoring | Social Support Group
Number analyzed (Participants) | 122 | 129
units on a scale | 33.16 (0.40) | 33.12 (0.39)

3. Secondary Outcome: Treatment Credibility
Description: To assess for differences in outcome expectancy, a modified treatment credibility scale developed by Borkovec and Nau (1972) will be used. Four of the questions will be used for this study, with 10-point Likert scales. These include questions regarding how logical the treatment seems, how confident participants are about treatment, and their expectancy of success
Time Frame: Baseline to 12 months post-intervention
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Satisfaction With Care: Validated General Scale
Description: Satisfaction with Care will be measured with a previously validated general scale to measure satisfaction/dissatisfaction with health care. The 2-item scale ranges from 1 (Strongly Agree) to 5 (Strongly Disagree).
Time Frame: Baseline to 12 months post-intervention
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Disease Activity Measured by the Systemic Lupus Activity Questionnaire (SLAQ)
Description: The Systemic Lupus Activity Questionnaire (SLAQ) asks a single Patient Global Assessment (PGA) question about presence and severity of lupus activity over the past month, questions on 24 specific symptoms of disease activity and a single Numerical Rating Scale (NRS) asking the patient to rate disease activity on a scale of 0-10 over the past three months. The reported patient global assessment has a scale of 0-3. A higher score represents a better outcome.
Time Frame: Baseline to 12 months post-intervention
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Mentoring | Social Support Group
Number analyzed (Participants) | 122 | 129
units on a scale | 1.13 (0.08) | 1.19 (0.08)

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Peer Mentoring: Peer Mentors: Peer mentors administered the peer mentoring intervention and were not involved in social support groups.
Arm/Group | Peer Mentoring | Social Support Group | Peer Mentoring: Peer Mentors
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/129 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/129 | 0/44
Other Adverse Events (participants affected / at risk) | 0/122 | 0/129 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT03734055/Prot_SAP_000.pdf